CLINICAL TRIAL: NCT06031389
Title: Henagliflozin Delays the Progress of Diabetic Nephropathy Via Regulates Gut-Renal Axis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Zunsong Wang, Director, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HENA-DKD
Record Dates: First submitted 2023-07-29; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Nephropathies
Keywords: Henagliflozin; Diabetic Nephropathy; enteric microorganisms
MeSH Terms: conditions — Diabetic Nephropathies | interventions — henagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Henagliflozin (Experimental): On the basis of basic treatment, the patients in the Hengglinide（tabuletta） intervention group were given Hengglinide once a day, 10mg or 5mg each time in the morning, and continued to intervene for 12 months.
  Interventions: Drug: Henagliflozin
- Placebo (Placebo Comparator): The blank control group was treated with placebo (starch tablets) once a day, 10mg or 5mg each time, taken in the morning for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Henagliflozin — On the basis of hypoglycemic therapy, the patients in the intervention group were given the drug treatment of hengglinide, once a day, 10mg or 5mg each time, taken in the morning, for 12 months.
  Arms: Henagliflozin
Drug: Placebo — On the basis of basic treatment, patients in the blank control group were given starch tablets once a day, 10mg or 5mg each time, taken in the morning for 12 months.
  Arms: Placebo

SUMMARY:
Diabetic kidney disease (DKD) is a serious complication of diabetes, and it is also the leading cause of end-stage renal disease (ESRD) in the world. The aggravation of progressive proteinuria and the decrease of glomerular filtration rate are the important reasons for the development of DKD into ESRD. It is an important task in the medical field to delay the development of DKD into ESRD. In recent years, gut microbiota disorder has been considered as an important influencing factor of DKD, and the concept of gut-renal axis has attracted more and more attention. The disorder of gut microbiota in DKD patients is mainly manifested by the decrease in the abundance of probiotics such as Lactobacillus, Bifidobacterium and Akkermansia, which produce short-chain fatty acids (SCFA), and the increase in the abundance of uremic toxin-producing bacteria such as Ruminococcus, Alistipes and Subdoligranulum. Improving gut microbiota disorder and increasing the concentration of beneficial metabolites such as SCFA in serum have positive effects on improving DKD. In recent years, with the application of sodium-glucose cotransporter 2 inhibitors (SGLT-2i), diabetes has been effectively treated. SGLT-2i can reduce blood glucose concentration by inhibiting renal tubular glucose reabsorption, and at the same time, it can play a renal protection role independent of blood glucose reduction by correcting the unbalanced tubuloglomerular feedback during diabetes and improving inflammation. However, the mechanism of its renal protection seems to be more than that. Studies have shown that SGLT-2i can reduce proteinuria in DKD mice by regulating the disordered gut microbiota during DKD, but not all SGLT-2i preparations have the effect of protecting target organs by regulating gut microbiota. Wang found that canagliflozin can regulate the gut microbiota of diabetes mice and improve cardiovascular complications; Lee reported that dapagliflozin could reduce the ratio of Firmicutes/Bacteroides in DKD mice and increase the abundance of Akkermansia. Yang found that dapagliflozin increased the abundance of Proteobacteria in diabetes rats, but it did not seem to affect the ratio of Firmicutes/Bacteroides. Van Bommel reported that dapagliflozin would not affect the gut microbiot of diabetes patients. Whether henagliflozin can improve DKD by regulating the gut-renal axis is worthy of further study.

ELIGIBILITY:
Inclusion Criteria:

1.18-65 years old, regardless of gender; 2. It was confirmed as DKD by renal biopsy. 3. It needs to be treated with DKD standard scheme, but it can be adjusted according to needs.

4.eGFR>30ml/min/1.73m2 5.200mg/g<UACR<5000mg/g 6. Stabilize the maximum tolerated dose ACEi/ARB ≥4 weeks. 7. Volunteer to participate in the study, understand the significance of this experiment and the indicators to be measured, and sign the informed consent form.

Exclusion Criteria:

1. Severe infection: there are clinical manifestations such as fever, cough and expectoration, sore throat, abdominal pain, diarrhea, carbuncle and furuncle, and the white blood cell count in blood is beyond the normal range (10× 109/L); 2. Severe hypoproteinemia (albumin < 20g/L) 3 malnutrition or BMI<18.5 kg/m2. 4. Hemoglobin < 60g/L; 5. No full capacity; 6. Severe hypotension (< 90/60mmhg); 7. Severe hypertension (> 180/110mmHg). Have used SGLT2i of any kind, dosage and dosage form within 8.6 months or are intolerant of such drugs.

9.1 type diabetes mellitus 10. Patients who have had ketoacidosis, diabetic coma or multiple hypoglycemia episodes in the past.

11. Polycystic kidney disease, lupus nephritis, ANCA- related vasculitis. 12. Immunosuppressant treatment for 6 months or less before enrollment. 13. Severe heart failure (NYHA grade ≧II-III) 14. Other serious heart diseases, such as recent myocardial infarction, persistent atrial fibrillation and valvular heart disease.

15 patients with severe liver dysfunction (ALT or AST>3 times the normal upper limit, or total bilirubin > 2 times the normal upper limit) 16. Chronic cystitis, or urinary tract infection ≥3 times within 1 year. 17 patients with obvious bleeding tendency or blood system diseases, or patients with bone marrow suppression.

18. Malignant tumor 19. Pregnant women, lactating patients or patients who plan to become pregnant. 20. There are acute or severe systemic infections. 21. The subject is participating in clinical trials of other drugs or medical devices.

22. Any known drug or alcohol dependence, difficulty in understanding the trial protocol, and inability or unwillingness to follow up according to the trial protocol.

23. Moderate and severe cognitive impairment and no long-term fixed guardian. 24. Chronic diarrhea and indigestion 25. Patients that the researcher thinks are not suitable to participate in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of intestinal flora difference between intervention group and control group with diabetic nephropathy by bacterial 16srDNA sequencing | baseline、1 month、3 month、6 month and 12 month
  16srDNA sequencing was used to detect the difference of relative abundance of different kinds of intestinal flora between the two groups.

SECONDARY OUTCOMES:
Statistical analysis of the degree of proteinuria relief in intervention group and control group. | baseline、1 month、3 month、6 month and 12 month
  T-test or Wilcoxon rank-sum test were used to compare the difference of urinary microalbumin creatinine ratio in two groups of diabetic nephropathy patients in regular urine biochemical tests.